CLINICAL TRIAL: NCT00491829
Title: A Twenty-Four Week, Randomized, Double-Blind, Placebo Controlled, Safety and Efficacy Trial of Flibanserin 50 Milligrams Daily and 100 Milligrams Daily in Premenopausal European Women With Hypoactive Sexual Desire Disorder
Brief Title: Flibanserin Versus Placebo in Premenopausal Women With HSDD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sprout Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 511.77
Record Dates: First submitted 2007-06-25; First posted 2007-06-26 (Estimated); Results first posted 2014-06-02 (Estimated); Last update posted 2014-06-02 (Estimated); Status verified 2014-05

CONDITIONS: Sexual Dysfunctions, Psychological
MeSH Terms: conditions — Sexual Dysfunctions, Psychological

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- flibanserin (Experimental): 50 mg qhs
  Interventions: Drug: 50 mg qhs
- flibanserin 100mg (Experimental): 100 mg qhs
  Interventions: Drug: 100 mg
- placebo (Placebo Comparator): placebo qhs
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: 50 mg qhs — flibanserin 50 mg
  Arms: flibanserin
Drug: 100 mg — flibanserin 100mg
  Arms: flibanserin 100mg
Drug: placebo — placebo
  Arms: placebo

SUMMARY:
To establish efficacy of Flibanserin 50 Milligrams Daily and 100 Milligrams Daily in 6-month treatment, vs placebo for Hypoactive Sexual Desire Disorder in premenopausal European women.

To evaluate safety and tolerability of flibanserin in such patients.

ELIGIBILITY:
Inclusion Criteria:

1. Women who are 18 years of age and older at the Screen Visit.
2. Premenopausal women per the Stages of Reproductive Aging Workshop (STRAW) criteria with the primary diagnosis of HSDD, generalized acquired type, according to DSM IV-TR criteria. The current episode must be at least 24 weeks in duration by the Baseline Visit. Secondary Female Sexual Arousal Disorder and/or Female Orgasmic Disorder are allowed. This inclusion criterion is met only if the HSDD commenced prior to Female Sexual Arousal Disorder and/or Female Orgasmic Disorder and the HSDD is of more importance to the patient, in the investigator judgement
3. A score of 15 or higher on the Female Sexual Distress Scale-Revised (FSDS-R)© (R04-1068) at the Screen Visit.
4. Item Number Two of the Sexual Interest and Desire Inventory - Female© (SIDI-F©) must be rated as "0" or "1" at the Screen Visit
5. Patients must be willing to try to have sexual activity (e.g., any act involving direct genital stimulation) at least once monthly.
6. Patients must be willing and able to use an eDiary on a daily basis (e.g., have access to a working land line or wireless telephone for daily data transmissions).
7. At the Baseline Visit, patients must have complied with eDiary use adequately, having missing entries for five or less days during the 28-day Screen period.
8. Patients must be in a stable, monogamous, heterosexual relationship that is secure and communicative, for at least 1 year prior to the Screen Visit. The relationship is to be with the same partner who is sexually functional, both psychologically and physically, and the partner is expected to be physically present (i.e., available for sexual activity at some time during a 24 hour day) at least 50% of each month during the 4-week Screen period and 24-week efficacy period of the trial.

Exclusion Criteria:

1. Patients who have taken any medication noted in Appendix 10.6.1, Part I - List of prohibited medications, within 30 days before the Screen Visit; the same medications are prohibited throughout participation in the study.
2. Patients whose sexual function was affected (enhanced or worsened) in the investigator opinion by any medication within 30 days before the Screen Visit and anytime prior to the Baseline Visit. This must be determined by the investigator judgement after performing a detailed review of the patient sexual history and concomitant therapy.
3. Patients with a history of drug dependence or abuse (including alcohol, as defined in DSM IV-TR or in the opinion of the investigator) within the past 1 year
4. Patients who meet DSM IV-TR criteria for Sexual Aversion Disorder, Substance-Induced Sexual Dysfunction, Dyspareunia (not caused by inadequate foreplay stimulation or alleviated by lubricants), Vaginismus, Gender Identity Disorder, Paraphilia, or for Sexual Dysfunction Due to a General Medical Condition.
5. Patients who indicate that their sexual partner has organic or psychosexual dysfunction that could interfere with a patient response to treatment.
6. Patients who have entered the peri-menopause stage (menopausal transition) or the post menopause stage [i.e., have had hysterectomy (without bilateral oophorectomy), bilateral oophorectomy, endometrial ablation (any type), and chemical induced (e.g., chemotherapy)] according to the STRAW criteria.
7. Patients with a history of MDD within 6 months prior the Screen Visit or a score of 14 on the Beck Depression Inventory© II, or a history of suicide attempt according to the Beck Scale for Suicide Ideation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 945 (Actual)
Dates: Start 2007-06; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (86):
- Austria (5):
  - 511.77.43005 Boehringer Ingelheim Investigational Site, Innsbruck
  - 511.77.43001 Boehringer Ingelheim Investigational Site, Vienna
  - 511.77.43002 Boehringer Ingelheim Investigational Site, Vienna
  - 511.77.43004 Boehringer Ingelheim Investigational Site, Vienna
  - 511.77.43006 Boehringer Ingelheim Investigational Site, Wörgl
- Belgium (5):
  - 511.77.32004 Boehringer Ingelheim Investigational Site, Braine-l'Alleud
  - 511.77.32003 Boehringer Ingelheim Investigational Site, Edegem
  - 511.77.32005 Boehringer Ingelheim Investigational Site, Ghent
  - 511.77.32006 Boehringer Ingelheim Investigational Site, Hasselt
  - 511.77.32002 Boehringer Ingelheim Investigational Site, Yvoir
- Czechia (4):
  - 511.77.42001 Boehringer Ingelheim Investigational Site, Olomouc
  - 511.77.42002 Boehringer Ingelheim Investigational Site, Prague
  - 511.77.42003 Boehringer Ingelheim Investigational Site, Prague
  - 511.77.42004 Boehringer Ingelheim Investigational Site, Vřesina
- Finland (5):
  - 511.77.35801 Boehringer Ingelheim Investigational Site, Espoo
  - 511.77.35805 Boehringer Ingelheim Investigational Site, Helsinki
  - 511.77.35802 Boehringer Ingelheim Investigational Site, Oulu
  - 511.77.35803 Boehringer Ingelheim Investigational Site, Seinäjoki
  - 511.77.35804 Boehringer Ingelheim Investigational Site, Tampere
- France (13):
  - 511.77.3308A Boehringer Ingelheim Investigational Site, Blanquefort
  - 511.77.3301A Boehringer Ingelheim Investigational Site, Bordeaux
  - 511.77.3305A Boehringer Ingelheim Investigational Site, La Rochelle
  - 511.77.3314A Boehringer Ingelheim Investigational Site, Lille
  - 511.77.3314B Cabinet médical, Lille
  - 511.77.3314C Cabinet médical, Lille
  - 511.77.3303A Boehringer Ingelheim Investigational Site, Marseille
  - 511.77.3310A Boehringer Ingelheim Investigational Site, Marseille
  - 511.77.3312A Boehringer Ingelheim Investigational Site, Marseille
  - 511.77.3302A Boehringer Ingelheim Investigational Site, Paris
  - 511.77.3315A Cabinet Médical, Rennes
  - 511.77.3306A Boehringer Ingelheim Investigational Site, Saint-Émilion
  - 511.77.3311A Boehringer Ingelheim Investigational Site, Toulouse
- Germany (9):
  - 511.77.49004 Boehringer Ingelheim Investigational Site, Berlin
  - 511.77.49007 Boehringer Ingelheim Investigational Site, Bochum
  - 511.77.49001 Boehringer Ingelheim Investigational Site, Bonn
  - 511.77.49006 Boehringer Ingelheim Investigational Site, Dresden
  - 511.77.49008 Boehringer Ingelheim Investigational Site, Frankfurt
  - 511.77.49003 Boehringer Ingelheim Investigational Site, Freiburg im Breisgau
  - 511.77.49002 Boehringer Ingelheim Investigational Site, Hanover
  - 511.77.49005 Boehringer Ingelheim Investigational Site, Leipzig
  - 511.77.49009 Boehringer Ingelheim Investigational Site, Magdeburg
- Hungary (4):
  - 511.77.36001 Boehringer Ingelheim Investigational Site, Budapest
  - 511.77.36005 Boehringer Ingelheim Investigational Site, Kecskemét
  - 511.77.36003 Boehringer Ingelheim Investigational Site, Szeged
  - 511.77.36004 Boehringer Ingelheim Investigational Site, Szentes
- Italy (4):
  - 511.77.39004 Ospedale S. Bambino, Catania
  - 511.77.39001 IRCCS S. Fondazione Maugeri, Pavia
  - 511.77.39002 Ospedale Santa Chiara, Pisa
  - 511.77.39003 Ospedale Sant'Anna, Torino
- Netherlands (9):
  - 511.77.31006 Boehringer Ingelheim Investigational Site, Almere Stad
  - 511.77.31001 Boehringer Ingelheim Investigational Site, Amsterdam
  - 511.77.31004 Boehringer Ingelheim Investigational Site, Apeldoorn
  - 511.77.31007 Boehringer Ingelheim Investigational Site, Den Helder
  - 511.77.31005 Boehringer Ingelheim Investigational Site, Enschede
  - 511.77.31002 St Antonius ziekenhuis, Nieuwegein
  - 511.77.31009 Boehringer Ingelheim Investigational Site, The Hague
  - 511.77.31008 Boehringer Ingelheim Investigational Site, Tilburg
  - 511.77.31003 Boehringer Ingelheim Investigational Site, Zeist
- Norway (4):
  - 511.77.47002 Boehringer Ingelheim Investigational Site, Lillestrøm
  - 511.77.47001 Boehringer Ingelheim Investigational Site, Oslo
  - 511.77.47003 Boehringer Ingelheim Investigational Site, Oslo
  - 511.77.47004 Boehringer Ingelheim Investigational Site, Oslo
- Spain (6):
  - 511.77.34004 Boehringer Ingelheim Investigational Site, Barcelona
  - 511.77.34005 Boehringer Ingelheim Investigational Site, Barcelona
  - 511.77.34006 Boehringer Ingelheim Investigational Site, L´Hospitalet Del LLobregat
  - 511.77.34003 Boehringer Ingelheim Investigational Site, Manresa (Barcelona)
  - 511.77.34002 Boehringer Ingelheim Investigational Site, Mataró-Barcelona
  - 511.77.34001 Boehringer Ingelheim Investigational Site, Ourense
- Sweden (8):
  - 511.77.46004 Boehringer Ingelheim Investigational Site, Kungsbacka
  - 511.77.46009 Boehringer Ingelheim Investigational Site, Lund
  - 511.77.46007 Boehringer Ingelheim Investigational Site, Malmo
  - 511.77.46001 Junoenheten/Kvinnohälsan, Kvinnokliniken, Stockholm
  - 511.77.46002 Boehringer Ingelheim Investigational Site, Stockholm
  - 511.77.46006 Boehringer Ingelheim Investigational Site, Stockholm
  - 511.77.46005 Boehringer Ingelheim Investigational Site, Uppsala
  - 511.77.46003 Boehringer Ingelheim Investigational Site, Västerås
- United Kingdom (10):
  - 511.77.44011 Boehringer Ingelheim Investigational Site, Belfast
  - 511.77.44009 Boehringer Ingelheim Investigational Site, Chorley
  - 511.77.44004 Boehringer Ingelheim Investigational Site, Fisherwick, Lichfield
  - 511.77.44008 Boehringer Ingelheim Investigational Site, Glasgow
  - 511.77.44003 Boehringer Ingelheim Investigational Site, Headington, Oxford
  - 511.77.44005 Boehringer Ingelheim Investigational Site, Leeds
  - 511.77.44001 Boehringer Ingelheim Investigational Site, London
  - 511.77.44002 Boehringer Ingelheim Investigational Site, London
  - 511.77.44007 Boehringer Ingelheim Investigational Site, South Brent
  - 511.77.44010 Boehringer Ingelheim Investigational Site, Waterloo, Liverpool

RESULTS

PARTICIPANT FLOW:
Groups:
- Flibanserin 50mg: 50 mg qhs
  BIMT 17 BS 50 mg: flibanserin 50 mg
- Flibanserin 100mg: 100 mg qhs
  BIMT 17 BS 100 mg: flibanserin 100mg
Period: Overall Study
Arm/Group | Flibanserin 50mg | Flibanserin 100mg | Placebo
Started | 311 | 316 | 318
Completed | 216 | 202 | 243
Not Completed | 95 | 114 | 75

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Flibanserin 50mg | Flibanserin 100mg | Placebo | Total
Number analyzed (Participants) | 311 | 316 | 318 | 945
Age, Customized [Number; unit: participants]
  18-34 years | 145 | 128 | 148 | 421
  35-44 years | 133 | 157 | 147 | 437
  45 years and older | 33 | 31 | 23 | 87
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 311 | 316 | 318 | 945
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 276 | 281 | 286 | 843
  White Hispanic | 6 | 9 | 3 | 18
  Black | 2 | 3 | 3 | 8
  Black Hispanic | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 0 | 2
  Asian Hispanic | 0 | 0 | 0 | 0
  Missing | 26 | 22 | 26 | 74
Region of Enrollment [Number; unit: participants]
  Finland | 18 | 17 | 18 | 53
  Spain | 5 | 8 | 2 | 15
  Austria | 16 | 20 | 19 | 55
  Italy | 10 | 9 | 10 | 29
  United Kingdom | 31 | 34 | 35 | 100
  France | 27 | 27 | 28 | 82
  Hungary | 19 | 18 | 18 | 55
  Czech Republic | 22 | 20 | 21 | 63
  Belgium | 27 | 27 | 28 | 82
  Netherlands | 30 | 32 | 34 | 96
  Norway | 11 | 13 | 10 | 34
  Germany | 56 | 54 | 55 | 165
  Sweden | 39 | 37 | 40 | 116

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Frequency of Satisfying Sexual Events as Measured by the eDiary.
Description: To obtain information on satisfying sexual events (SSEs), a small personal handheld electronic device was to be used by the patients to record such information daily (eDiary). An SSE was recorded when a patient answered "yes" to the eDiary question: "Was the event satisfying for you?"
Time Frame: baseline to 24 weeks
Population: Patients who had at least one post-dose on-treatment efficacy assessment were included in the Full Analysis Set (FAS). The FAS was used for primary analyses.
Measure: Mean (Standard Deviation); unit: events per month
Arm/Group | Flibanserin 50mg | Flibanserin 100mg | Placebo
Number analyzed (Participants) | 297 | 299 | 307
events per month | 1.2 (3.7) | 1.5 (4.0) | 0.9 (3.2)

ADVERSE EVENTS:
Arm/Group | Flibanserin 50mg | Flibanserin 100mg | Placebo
Serious Adverse Events (participants affected / at risk) | 25/311 | 19/316 | 16/318
Other Adverse Events (participants affected / at risk) | 174/311 | 238/316 | 143/318
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Flibanserin 50mg (N=311) | Flibanserin 100mg (N=316) | Placebo (N=318)
haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
ovarian cyst ruptured (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 0 (0)
abdominal pain (Gastrointestinal disorders) | 9 (12) | 6 (6) | 6 (6)
gliosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
metrorrhagia (Reproductive system and breast disorders) | 12 (14) | 9 (13) | 6 (9)
suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
subileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
circulatory collapse (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
concussion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Flibanserin 50mg (N=311) | Flibanserin 100mg (N=316) | Placebo (N=318)
Headache (Nervous system disorders) | 49 (91) | 53 (66) | 42 (67)
Dizziness (Nervous system disorders) | 23 (25) | 46 (55) | 14 (16)
Somnolence (Nervous system disorders) | 12 (12) | 16 (17) | 3 (3)
nasopharyngitis (Infections and infestations) | 36 (45) | 30 (35) | 32 (37)
nausea (Gastrointestinal disorders) | 19 (20) | 39 (49) | 19 (20)
Fatigue (General disorders) | 35 (41) | 54 (67) | 33 (36)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No